CLINICAL TRIAL: NCT00534391
Title: Dose Antibiotic Need in Hordeolum After Incision and Curettage? : A Randomized, Placebo-controlled Trial
Brief Title: Comparison of Combination Antibiotics Eyedrop to Artificial Tear in Hordeolum After Incision and Curettage
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Department of Opthalmology, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 59/50
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Hordeolum
Keywords: Antibiotics; hordeolum
MeSH Terms: conditions — Hordeolum | interventions — Neomycin; Polymyxin B; Gramicidin; bacitracin zinc, neomycin sulfate, polymyxin B, drug combination; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (Placebo Comparator): Artificial tear containing antibiotic solution base
  Interventions: Drug: Artificial tear
- A (Experimental): combined antibiotic ophthalmic solution (neomycin sulfate, polymyxin B sulfate and gramicidin)
  Interventions: Drug: neomycin sulfate, polymyxin B sulfate and gramicidin

INTERVENTIONS:
Drug: neomycin sulfate, polymyxin B sulfate and gramicidin — to the effected eye 4 times a day
  Other Names: Neosporin; Polyoph
  Arms: A
Drug: Artificial tear — 4 times daily
  Other Names: Tear natural II; Lacoph
  Arms: B

SUMMARY:
To compare the effectiveness of combined antibiotic ophthalmic solution (neomycin sulfate, polymyxin B sulfate and gramicidin) with placebo (artificial tear) in the treatment of hordeolum after incision and curettage

DETAILED DESCRIPTION:
Hordeolum is a common eyelid disease. In case of mass, I&C is required but role of antibiotic after I&C is not clear. It may not need in post drainage period.

ELIGIBILITY:
Inclusion Criteria:

* at least 5-millimeters hordeolum
* the onset within 7 days

Exclusion Criteria:

* previous incision and curettage of the same site within 1 month or more than 3 times
* lesions in the adjacent areas suggesting of complications associated with hordeolum such as preseptal cellulitis or blepharitis
* The patients with immunodeficiency, history of bleeding tendency
* allergy to aminoglycoside, polymyxin B, gramicidin, xylocaine and povidone iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-09; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pain scale | 1,3,7 days after treatment

SECONDARY OUTCOMES:
Mass size and duration of cure | 1, 3, 7, 30 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Parima Hirunwiwatkul, MD, Principal Investigator — Department of Ophthalmology, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Department of Ophthalmology, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Background] Hirunwiwatkul P, Wachirasereechai K. Effectiveness of combined antibiotic ophthalmic solution in the treatment of hordeolum after incision and curettage: a randomized, placebo-controlled trial: a pilot study. J Med Assoc Thai. 2005 May;88(5):647-50. PMID 16149682